CLINICAL TRIAL: NCT06245733
Title: Investigation of the Effect of Compassion-Based Education Program Applied to the Mothers of Children Diagnosed With Cerebral Palsy on Compassion, Depression and Resilience
Brief Title: Study of the Effect of Compassion-Based Education Program Applied to Mothers of Children Diagnosed With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat SEVEN, Director, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MSEVEN
Record Dates: First submitted 2023-08-02; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
Keywords: Serebral Palsi; Depression; Resilience; Compassion
MeSH Terms: conditions — Cerebral Palsy; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants who will receive the training
  Interventions: Other: Compassion-Based Education Program Adapted for Adults
- Control Group (No Intervention): participants who will not be interfered with

INTERVENTIONS:
Other: Compassion-Based Education Program Adapted for Adults — Training will be given once a week. This training will last 10 weeks in total.
  Arms: Experimental Group

SUMMARY:
Purpose of the study; The aim of this study is to examine the effect of a compassion-based education program applied to mothers of children with cerebral palsy on compassion fatigue, depression, and psychological resilience.

DETAILED DESCRIPTION:
The Hypotheses of the Study

Main Hypothesis: "Compassion-Based Education Program Adapted for Adults" in increasing the compassion levels and psychological resilience of mothers of patients with CP; It is effective in reducing the level of depression.

As sub-hypotheses:

H1: The scores of the mothers who care for their children with Cerebral Palsy in the experimental group at the end of the application (post-test) and after the application (follow-up test) of the Adult Compassion Scale are significantly higher than the scores they obtained before the application (pre-test).

H2: The scores of the mothers who care for their children with Cerebral Palsy in the experimental group at the end of the application (post-test) and after the application (follow-up test) of the Burns Depression Scale-Turkish Form are significantly lower than the scores they obtained before the application (pre-test).

H3: The scores of the mothers who care for their children with Cerebral Palsy in the experimental group at the end of the application (post-test) and after the application (follow-up test) of the Adult Resilience Scale are significantly higher than the scores they obtained before the application (pre-test).

ELIGIBILITY:
Inclusion Criteria:

* Being the mother of a child with Cerebral Palsy

Exclusion Criteria:

* Mothers who have children with Cerebral Palsy do not want to participate in the study and want to leave the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment and Evaluation of Depression | Day 1
  Burns Depression Scale will be applied to all participants. Depression levels will be determined.
Assessment and Evaluation of Psychological Resilience | Day 1
  Psychological Resilience Scale for Adults will be applied to all participants. Psychological Resilience levels will be determined.
Assessment and Evaluation of Compassion | Day 1
  Compassion Scale will be applied to all participants. Compassion levels will be determined .

SECONDARY OUTCOMES:
The last test of Assessment and Evaluation of Depression | through study completion, an average of 1 week.
  Burns Depression Scale will be applied to all participants. Depression levels will be determined due to showing effectiveness of training.
The last test of Assessment and Evaluation of Psychological Resilience | through study completion, an average of 1 week.
  Psychological Resilience Scale will be applied to all participants. Resilience levels will be determined due to showing effectiveness of training.
The last test of Assessment and Evaluation Compassion | through study completion, an average of 1 week.
  Compassion Scale will be applied to all participants. Compassion levels will be determined due to showing effectiveness of training.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No